CLINICAL TRIAL: NCT01781260
Title: The Effect of Prone Positioning During Anaesthesia on Liver Blood Flow and Function
Brief Title: Effect of Prone Position on Liver Blood Flow and Function
Acronym: PLiF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 12098
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Prone Position; Cardiac Output; Liver Circulation
Keywords: Prone position; Cardiac output; Liver Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young. Fit. Minor neurosurgical operation. Prone position.: 18-65 year old patients, without serious medical co-morbidities (assessed as ASA I/II status) who are having minor to moderate severity neurosurgical operations in the prone position.

SUMMARY:
Recent occurrence of significant post-operative liver impairment at Nottingham University Hospitals NHS Trust has prompted investigation into whether interaction between general anaesthesia and prone positioning (lying face down) for surgery can influence liver function.

Historical research has shown that the heart does not function as efficiently when an anaesthetised patient is placed in the prone position for surgery. The techniques used for anaesthetising and monitoring these patients have changed remarkably, since these studies were first performed.

It is important to know accurately how the heart functions to enable better understanding of the changes in blood flow to the liver when in the prone position.

Studies looking at blood flow to the liver when lying face down have been done before but are mainly reporting patients on the intensive care unit. These intensive care patients are different to those in theatre undergoing routine surgery. The intensive care patients are usually received in different types of drugs and monitored with several different types of monitor at the time. Perhaps most importantly is that they are placed face down on a soft air cushioned mattress and pillows rather than the rigid support used for surgical patients.

This study will look at whether the function of the liver changes when a patient is anaesthetised and is then rolled onto their front. The function of the liver will be measured by looking how it clears a specific drug from the blood. Also this study will look at how accurate a particular type of heart monitor is when an anaesthetised patient is placed onto their front.

DETAILED DESCRIPTION:
Recent occurrence of significant post-operative hepatic dysfunction including two fatalities at Nottingham University Hospitals NHS Trust has prompted investigation into whether interaction between general anaesthesia, prone positioning for surgery, cardiac output and the use of vasoactive drugs can influence hepatic function.

Research has shown that cardiac output is decreased when an anaesthetised patient is placed from the supine to the prone position, and that the magnitude of these changes vary with the exact method of physical patient support in the prone position.1-3 Anaesthetic technique and methods of cardiac output monitoring used in these studies are no longer in routine use and therefore may not accurately reflect current practice of balanced anaesthesia or current monitoring techniques.

The LiDCOplus minimally invasive cardiac output monitor can be used to accurately calculate cardiac ouput and its associated derived variables (stroke volume and systemic vascular resistance). The LiDCOplus monitor uses data already available from an arterial cannula which is routinely used for monitoring patients in these circumstances. It is calibrated by using a small (0.3mmol) bolus dose of lithium chloride. This technique has been shown to be accurate and safe even after repeated calibration procedures over a short time period.4-6

Much of the evidence with regards to liver blood flow in the anaesthetised patient in prone position is from the critical care literature. There are several differences between this group of critically ill patients undergoing prone positioning for rescue therapy from refractory hypoxia due to acute lung injury and healthy patients undergoing elective surgery in the prone position. Critically ill patients have multiple cardiovascular and respiratory co-morbidities, are usually receiving infusions of vasoactive drugs and are generally positioned on soft air cushioned mattresses and pillows. Prone positioning in these patients does not seem to significantly alter hepatic function as measured by hepatic Indocyanine Green (ICG) clearance.7 8

ICG is a fluorescent dye, which can absorb infra-red light with a very rare (1:40 000) side effect profile. After intravenous injection it is almost exclusively eliminated by hepatic excretion into bile. The rate of hepatic elimination has been shown to correlate accurately with plasma disappearance rate as measured by transcutaneous infra-red absorbtion.9 It is a dynamic marker of hepatic blood flow, hepatocellular function and biliary excretion, with short term variation thought to be attributable to changes in hepatic blood flow rather than cellular dysfunction.10

The LiMON monitor uses transcutaneous infra-red light absorption (like a pulse oximeter) to measure and calculate values for ICG plasma disappearance and its associated values such as clearance rate and plasma retention rate. The technique involves intravenous injection of a small (0.25mg/kg) bolus dose of ICG. This can be repeated up to 20 times per 24hr period.

It is postulated that simultaneously measuring changes in hepatic blood flow and cardiac output will allow us to gather greater understanding of the haemodynamic changes associated with the prone position in the anaesthetised patient using current routine monitoring modalities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* ASA (American Society of Anaesthesiologists) I/II
* Surgery in prone position
* Classification of surgery as minor / moderate severity

Exclusion Criteria:

* Inability to give consent to inclusion in trial
* Unable to speak or read English
* Age less than 18 years
* Age over 65 years
* Pregnancy
* Pre-existing hepatic dysfunction
* Taking oral lithium (interferes with LiDCOplus calibration factor)
* Severe valvular heart disease (reduced reliability of LiDCO measurements)
* Major severity surgery with predicted large blood loss or alteration in aortic root anatomy
* Intolerance including allergy to lithium, iodine or ICG
* Thyrotoxicosis
* Patients expected to require radio active iodine studies within one week of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the age of 18-65, presenting for neurosurgical procedures to the Queen's Medical Centre, Nottingham, England, UK.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Liver blood flow and function as measured by non-invasive determination of ICG excretion. | During operative anaesthesia on day 1
  To test the null hypothesis that hepatic blood flow or global hepatic function does not change in the prone position during anaesthesia and therefore the ICG elimination rate remains constant and is unaffected by anaesthesia or patient position.

SECONDARY OUTCOMES:
Validating LiDCO calibration between supine and prone positions | During operative anaesthesia on day 1 of study
  To test the null hypothesis that calibration factor for the LiDCOplus monitor as determined by lithium dilution is not affected by changing the patient from supine to prone position.
Evaluation of change in cardiac output on position change. | During surgical anaesthesia on day 1 of study
  To test the null hypothesis that cardiovascular parameters as measured by the LiDCOplus monitor are not affected by changing the patient from supine to prone position.
Validation of preload predictors in the prone position. | During surgical anaesthesia on day 1 of study
  To test the null hypothesis that the dynamic indices of preload retain their discriminatory ability to predict positive response following a fluid bolus when the patient is placed in the prone position.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Centre Campus, Nottingham University Hospitals NHS Trust., Nottingham, Nottinghamshire, United Kingdom